CLINICAL TRIAL: NCT03222960
Title: Improving Caries Risk Using Propolis-containing Versus Fluoride-containing Toothpastes in High Caries Risk Patients: Randomized Clinical Trial
Brief Title: Improving Caries Risk Using Propolis-containing Versus Fluoride-containing Toothpastes in High Caries Risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Fawzy Meselhy Maarek, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEBC-CU-2017-07-26
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis-containing toothpaste (Experimental): Assessment of caries risk for participants using Propolis-containing toothpaste before the treatment , after 3 months and 6 months follow up.
  Interventions: Drug: propolis-containing toothpaste
- Fluoride-containing toothpaste (Experimental): Assessment of caries risk for participants using Fluoride-containing toothpaste before the treatment , after 3 months and 6 months follow up.
  Interventions: Drug: Fluoride-containing toothpaste

INTERVENTIONS:
Drug: propolis-containing toothpaste — participants will use propolis-containing toothpaste for 6 months
  Other Names: Red seal propolis toothpaste
  Arms: Propolis-containing toothpaste
Drug: Fluoride-containing toothpaste — participants will use Fluoride-containing toothpaste for 6 months
  Other Names: colgate
  Arms: Fluoride-containing toothpaste

SUMMARY:
This study will be conducted to evaluate the effect of Propolis-containing toothpaste in comparison to Fluoride-containing Toothpaste by caries risk assessment in high caries risk patients.

DETAILED DESCRIPTION:
A total of 40 patients will be assigned in this study. Patients will be randomly divided into two groups according to type of Toothpaste (A) where group A1 patients will use propolis containing toothpaste twice daily while group A2 patients will use fluoride containing toothpaste twice daily as control with 20 patients in each group. Each group will be further divided into three groups according to caries risk assessment times (T) where T0 represents caries risk assessment of patients before application of propolis and fluoride toothpastes and T1 represents caries risk assessment of patients after three months of application of propolis and fluoride toothpastes, T2 represents caries risk assessment of patients after six months of application of propolis and fluoride toothpastes.

Both Propolis containing toothpaste and fluoride containing toothpaste will be placed in concealed tubes. The tubes will completely wrapped by plain white tape to conceal the formulation of toothpaste. Participants are given the tubes of toothpaste and soft brush with a coloured mark at 2 cm length of the bristle surface. The technique can be summarised in four steps:

1. 2 cm of the toothpaste will be squeezed over the wet toothbrush bristles
2. The upper and lower teeth will be brushed for 2 min;
3. After brushing, the remaining toothpaste foam and saliva "slurry" will be swished around the dentition with active movements of the cheeks, lips and tongue, forcing the slurry in between the teeth for about 20 seconds before expectorating the slurry
4. No post-brushing water rinsing will be carried out All these steps will be presented in a reminder card and all patients will put a tick mark for every step.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be over 18 years of age.
* Participants should be high caries risk.
* Systematically healthy.
* Not taking any medication interfering with saliva secretion.
* Participants who signed informed consent.

Exclusion criteria:

* Participants with a compromised medical history.
* Participants under systemic disease treatment, with antibiotic, steroid or any medication known to cause dry mouth.
* Severe or active periodontal disease.
* History of allergies or other adverse reactions to propolis, or oral care product or their ingredient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Improving caries risk | 6 months
  caries risk assessment